CLINICAL TRIAL: NCT00556374
Title: A Randomised, Double-Blind, Placebo-Controlled, Multi-Centre Phase 3 Study to Determine the Treatment Effect of Denosumab in Subjects With Non-Metastatic Breast Cancer Receiving Aromatase Inhibitor Therapy.
Brief Title: Study to Determine Treatment Effects of Denosumab in Patients With Breast Cancer Receiving Aromatase Inhibitor Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Austrian Breast and Colorectal Cancer Study Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20050209; ABCSG-18 (Other: Austrian Breast and Colorectal Cancer Study Group); 2005-005275-15 (EudraCT Number)
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: confirmed adenocarcinoma; non-metastatic breast cancer; estrogen receptor positive; progesterone receptor positive; non-steroidal aromatase; aromatase inhibitor therapy; postmenopausal woman; adjuvant chemotherapy; neoadjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Denosumab; Zoledronic Acid; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Denosumab (Experimental): Participants received 60 mg denosumab subcutaneous injection once every 6 months. All participants continued to receive an approved non-steroidal aromatase inhibitor therapy.
  Interventions: Biological: Denosumab; Drug: Non-steroidal aromatase inhibitor therapy
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injection once every 6 months. All participants continued to receive an approved non-steroidal aromatase inhibitor therapy.
  Interventions: Drug: Placebo; Drug: Non-steroidal aromatase inhibitor therapy
- SubStudy: Zoledronic Acid (Experimental): Eligible participants who completed the open-label phase could be enrolled into the zoledronic acid substudy and randomized to receive a single 5 mg intravenous dose of zoledronic acid 8 months after the last open-label dose of denosumab.
  Interventions: Drug: Zoledronic Acid
- Substudy: Standard of Care (Other): Eligible participants who completed the open-label phase could be enrolled into the zoledronic acid substudy and randomized to receive standard of care 8 months after the last open-label dose of denosumab.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Placebo
  Other Names: Administered as a subcutaneous injection
  Arms: Placebo
Biological: Denosumab — Administered as a subcutaneous injection
  Other Names: Prolia®
  Arms: Denosumab
Drug: Non-steroidal aromatase inhibitor therapy — An approved non-steroidal aromatase inhibitor therapy (eg, anastrazole) in the adjuvant setting
  Arms: Denosumab; Placebo
Drug: Zoledronic Acid — 5 mg zoledronic acid administered at a constant infusion rate
  Other Names: Reclast; Zometa
  Arms: SubStudy: Zoledronic Acid
Other: Standard of Care — Standard of care (SoC) as recommended by the treating physician, depending on individual factors such as bone density, lifestyle recommendations by the Investigator such as diet, physical activities and sun exposure, as well as local treatment standards.
  Arms: Substudy: Standard of Care

SUMMARY:
The purpose of this study is to determine whether denosumab compared to placebo, will reduce the rate of first clinical fracture in women with non-metastatic breast cancer receiving (non-steroidal) aromatase inhibitor therapy.

DETAILED DESCRIPTION:
Participants will remain on treatment until the required number of events (where an event is defined as first clinical fracture) is reached and all participants have had the opportunity to receive a minimum of at least 2 doses of study drug, whichever occurs later. The primary analysis data cut-off date (PADCD) is defined as the time at which the required number of events is reached and all participants have had the opportunity to receive at least 2 doses of study drug. When the PADCD is reached, all participants will discontinue study drug.

Following the study PADCD, participants will be followed every 12 months starting from their last study visit until a maximum of 66 months after PADCD.

After approval of Amendment 4, willing and eligible participants randomized to placebo during the double-blind phase may participate in an open-label phase (OLP) and receive denosumab 60 mg Q6M for up to 36 months (maximum of 7 doses).

After approval of Amendment 6 in 2019 a zoledronic acid (ZA) substudy was added to the protocol. Willing and eligible participants who participated in the OLP of the study and completed open-label denosumab may opt in to this ZA substudy and either receive a single dose of ZA (Therapy Arm), or be managed according to the current standard of care for this patient population (Control Arm).

ELIGIBILITY:
Inclusion Criteria for Double Blinded Phase:

* Histologically or cytologically confirmed adenocarcinoma of the breast;
* Female subjects with non-metastatic disease who are estrogen receptor (ER) and/or progesterone receptor (PR) positive, and who have completed their treatment pathway;
* Subjects who are currently on, or will initiate an approved non-steroidal aromatase inhibitor therapy (eg, anastrazole) in the adjuvant setting;
* Postmenopausal woman, defined as a woman fulfilling any one of the following criteria:

  * Having undergone a bilateral oophorectomy;
  * Age ≥ 60 years;
  * Aged < 60 years meeting the following requirements:
* Follicle-stimulating hormone (FSH) and estradiol in the postmenopausal range;
* A negative pregnancy test within 7 days prior to randomization. Subjects who have undergone a hysterectomy do not require a pregnancy test.
* More criteria may apply.

Exclusion Criteria for Double Blinded Phase:

* Aromatase inhibitor therapy for more than 24 months;
* Prior or concurrent treatment with Selective Estrogen Receptor Modulators (eg, tamoxifen);
* Evidence of metastatic disease;
* Current or prior intravenous (IV) bisphosphonate administration;
* Oral bisphosphonate treatment greater than or equal to 3 years continuously OR greater than 3 months but less than 3 years unless there was a washout period of at least 1 year prior to randomization OR any use during the 3-month period prior to randomization;
* Prior administration of denosumab;
* Known liver or renal deficiency;
* Recurrence of the primary malignancy (e.g., during the allowed interval of pretreatment with aromatase inhibitor);
* Diagnosis of any second non-breast malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or for in situ carcinoma of the cervix uteri;
* Any kind of disorder that compromises the ability to give written informed consent and/or comply with study procedures.

Inclusion Criteria to Receive Open-label Phase Denosumab:

* Obtain signed and dated written informed consent prior to performing any study-specific procedure;
* Subjects currently taking an approved non-steroidal AIT (eg, anastrazole) or who have completed or discontinued AIT within 12 months prior to participation in the OLP;
* Randomized to placebo arm during the double-blind phase (as determined by unblinding procedures);

Exclusion Criteria to Receive Open-label Phase Denosumab:

* Current or prior IV bisphosphonate administration;
* Subjects meeting the following criteria for oral bisphosphonate treatment:

  * Greater than or equal to 3 years continuously,
  * Greater than 3 months but less than 3 years unless subject has had a washout period of at least 1 year prior to participation in the OLP,
  * Any use during the 3-month period prior to participation in the OLP;
* Prior or concurrent treatment with SERMs (eg, tamoxifen);
* Subjects who ended treatment with investigational product (IP) prematurely in the double-blind phase; Treatment with commercial denosumab (Prolia or Xgeva) prior to participation in the OLP.

Eligibility for ZA substudy Inclusion Criteria

* Obtain signed and dated written informed consent prior to performing any substudy-specific procedure
* Subjects that received OLP denosumab and completed OLP treatment
* Last OLP denosumab administration no longer than 9 months ago Exclusion Criteria
* Current or prior ZA administration.
* Subjects who ended treatment with investigational product (IP) prematurely in the double-blind phase and OL phase
* Known sensitivity or intolerance to any of the products to be administered during the substudy (eg, ZA, calcium or vitamin D)
* Known history of any of the following conditions either by subject self report or chart review

  * Paget's disease (bone), Cushing's disease, hyperprolactinemia or other active metabolic bone disease
  * Known history of hypocalcemia
  * Major surgery, or significant traumatic injury occurring within 4 weeks prior to randomization
  * Parathyroid glands in neck surgically removed.
  * Any sections of intestine removed.
  * Known human immunodeficiency virus infection
  * Active infection with hepatitis B or hepatitis C virus
* Known liver or renal disease as determined by the investigator and indicated by the following criteria:

  * Aspartate aminotransferase ≥ 2.5 x ULN
  * Alanine transaminase ≥ 2.5 x ULN
  * Serum creatinine ≥ 2 x ULN
  * Creatine clearance < 35ml/min Subjects that are pregnant or breastfeeding
  * All subjects with reproductive potential must have a negative pregnancy test within 7 days before randomization
* Subjects who are osteoporotic in baseline BMD

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3420 (Actual)
Dates: Start 2006-12-18 (Actual); Primary Completion 2014-10-07 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (34):
- Austria (30):
  - Research Site, Baden
  - Research Site, Braunau am Inn
  - Research Site, Dornbirn
  - Research Site, Feldkirch
  - Research Site, Gmunden
  - Research Site, Graz
  - Research Site, Güssing
  - Research Site, Hall in Tirol
  - Research Site, Innsbruck
  - Research Site, Klagenfurt
  - Research Site, Krems
  - Research Site, Kufstein
  - Research Site, Leoben
  - Research Site, Lienz
  - Research Site, Linz
  - Research Site, Oberpullendorf
  - Research Site, Ried
  - Research Site, Rottenmann
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Sankt Veit an der Glan
  - Research Site, Schärding
  - Research Site, Steyr
  - Research Site, Vienna
  - Research Site, Villach
  - Research Site, Vöcklabruck
  - Research Site, Weiz
  - Research Site, Wels
  - Research Site, Wiener Neustadt
  - Research Site, Wolfsberg
- Sweden (4):
  - Research Site, Gävle
  - Research Site, Gothenburg
  - Research Site, Stockholm
  - Research Site, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Gnant M, Pfeiler G, Dubsky PC, Hubalek M, Greil R, Jakesz R, Wette V, Balic M, Haslbauer F, Melbinger E, Bjelic-Radisic V, Artner-Matuschek S, Fitzal F, Marth C, Sevelda P, Mlineritsch B, Steger GG, Manfreda D, Exner R, Egle D, Bergh J, Kainberger F, Talbot S, Warner D, Fesl C, Singer CF; Austrian Breast and Colorectal Cancer Study Group. Adjuvant denosumab in breast cancer (ABCSG-18): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet. 2015 Aug 1;386(9992):433-43. doi: 10.1016/S0140-6736(15)60995-3. Epub 2015 May 31. PMID 26040499
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Gnant M, Frantal S, Pfeiler G, Steger GG, Egle D, Greil R, Fitzal F, Wette V, Balic M, Haslbauer F, Melbinger-Zeinitzer E, Bjelic-Radisic V, Artner-Matuschek S, Kainberger F, Ritter M, Rinnerthaler G, Sevelda P, Bergh J, Kacerovsky-Strobl S, Suppan C, Brunner C, Deutschmann C, Gampenrieder SP, Fohler H, Jakesz R, Fesl C, Singer C. Long-Term Outcomes of Adjuvant Denosumab in Breast Cancer. NEJM Evid. 2022 Dec;1(12):EVIDoa2200162. doi: 10.1056/EVIDoa2200162. Epub 2022 Nov 18. PMID 38319865
- [Derived] Minichsdorfer C, Fuereder T, Leutner M, Singer CF, Kacerovsky-Strobl S, Egle D, Greil R, Balic M, Fitzal F, Pfeiler G, Frantal S, Bartsch R, Gnant M. Effect of concomitant statin treatment in postmenopausal patients with hormone receptor-positive early-stage breast cancer receiving adjuvant denosumab or placebo: a post hoc analysis of ABCSG-18. ESMO Open. 2022 Apr;7(2):100426. doi: 10.1016/j.esmoop.2022.100426. Epub 2022 Mar 22. PMID 35334418
- [Derived] Gnant M, Pfeiler G, Steger GG, Egle D, Greil R, Fitzal F, Wette V, Balic M, Haslbauer F, Melbinger-Zeinitzer E, Bjelic-Radisic V, Jakesz R, Marth C, Sevelda P, Mlineritsch B, Exner R, Fesl C, Frantal S, Singer CF; Austrian Breast and Colorectal Cancer Study Group. Adjuvant denosumab in postmenopausal patients with hormone receptor-positive breast cancer (ABCSG-18): disease-free survival results from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Mar;20(3):339-351. doi: 10.1016/S1470-2045(18)30862-3. Epub 2019 Feb 19. PMID 30795951
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 58 centers in Austria and Sweden from December 2006 to August 2020.
  Data collected during the exploratory ZA substudy were not used for the final analysis of the main study.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive either denosumab or placebo in the double-blind phase. Randomization was stratified by type of hospital (major academic centers or other centers), prior aromatase inhibitor usage (Yes/No) and total lumbar spine bone mineral density (BMD) score at baseline (T-score < -1.0 or ≥ -1.0). Willing and eligible participants continued into the open-label phase and receive denosumab for a maximum of 7 doses once Q6M.
Groups:
- Placebo: Participants randomized to receive the matching placebo subcutaneously (SC) once every 6 months (Q6M) in the double-blind phase. All participants continued to receive an approved non-steroidal aromatase inhibitor therapy.
- Denosumab: Participants randomized to receive 60 mg denosumab SC once Q6M in the double-blind phase. All participants continued to receive an approved non-steroidal aromatase inhibitor therapy.
Period: Overall Study
Arm/Group | Placebo | Denosumab
Started | 1709 | 1711
Received Study Drug in the Double-blind Phase | 1699 | 1700
Continued Into the Open-Label Phase | 268 | 3
Safety Analysis Set | 1690 (The safety analysis set was summarized based on the actual treatment received in the double-blind phase. Participants who received at least 1 dose of denosumab in the double-blind phase were summarized in the denosumab group regardless of the randomized treatment.) | 1709 (The safety analysis set was summarized based on the actual treatment received in the double-blind phase. Participants who received at least 1 dose of denosumab in the double-blind phase were summarized in the denosumab group regardless of the randomized treatment.)
Completed | 1242 | 1362
Not Completed | 467 | 349
Not completed — Withdrawal by Subject | 235 | 205
Not completed — Death | 158 | 127
Not completed — Lost to Follow-up | 24 | 17
Not completed — Continuing into Zoledronic Acid Substudy | 50 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab | Total
Number analyzed (Participants) | 1709 | 1711 | 3420
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (8.0) | 64.0 (7.9) | 64.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1709 | 1711 | 3420
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 1700 | 1702 | 3402
  Asian | 7 | 5 | 12
  Hispanic/Latino | 1 | 3 | 4
  Black/Afro-Caribbean | 0 | 1 | 1
  Missing | 1 | 0 | 1
Stratification Factor: Type of Hospital [Number; unit: participants]
  Major Academic Center | 632 | 633 | 1265
  Other Center | 1077 | 1078 | 2155
Stratification Factor: Prior Aromatase inhibitor Use [Count of Participants; unit: Participants]
  No | 269 | 270 | 539
  Yes | 1440 | 1441 | 2881
Stratification Factor: Total Lumbar Spine BMD T-score [Count of Participants; unit: Participants] — T-scores are standardized scores that reflect the standard deviations (SDs) above/below the normal mean for young adults.
  T-score ≥ -1.0: BMD is considered normal.
  T-score < -1.0: Low BMD.
  Participants
    T-score < -1.0 | 775 | 773 | 1548
    T-score ≥ -1.0 | 934 | 938 | 1872

OUTCOME MEASURES:

1. Primary Outcome: Time to First Clinical Fracture
Description: The time to first on-study clinical fracture was defined as the number of days from randomization to the date of the x-ray confirming the clinical fracture. A clinical fracture is any clinically evident fracture with associated symptoms and confirmed by x-ray. Participants who died or withdrew without experiencing a clinical fracture were censored at the date of last contact or study termination whichever was earlier.
Time Frame: From randomization until the primary analysis cut-off date of 26 March 2014; maximum time on main study at the cut-off was 87 months
Population: Full Analysis Set: all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 1709 | 1711
Days | NA [NA to NA] — Not reached due to the low number of events | NA [NA to NA] — Not reached due to the low number of events
Statistical Analysis 1: Comparison: Placebo vs Denosumab; The efficacy clinical hypothesis is that denosumab, when administered subcutaneously at a dose of 60 mg every 6 months, will be considered efficacious in patients with non-metastatic breast cancer receiving AIT if the rate of first clinical fracture in denosumab-treated patients is lower than that in placebo-treated patients. It is anticipated that denosumab will reduce the rate by 30% compared with placebo (ie, the true hazard ratio of denosumab compared with placebo is 0.70); Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazards Model; Stratification factors are hospital type, prior use of aromatase inhibitor, and baseline lumbar spine BMD; Hazard Ratio (HR) = 0.504, 95% CI 2-sided [0.39 to 0.65] — From the Cox proportional hazard model with treatment as the independent variable and stratified by randomization strata. A hazard ratio < 1.0 indicates a lower average event rate and a longer fracture-free time for denosumab relative to placebo

2. Secondary Outcome: Percent Change From Baseline in Total Lumbar Spine Bone Mineral Density (BMD) at Month 36 at Pre-selected Sites
Description: Bone mineral density was assessed by dual x-ray absorptiometry.
Time Frame: Baseline and Month 36
Population: BMD Analysis Set: all participants with evaluable lumbar spine BMD values at Baseline and Month 36
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change in BMD
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 245 | 230
Percent Change in BMD | -2.75 [-3.44 to -2.07] | 7.27 [6.56 to 7.98]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p < 0.0001, ANCOVA — The Hochberg procedure was used to control for multiplicity; Model includes treatment group as the independent variable and adjusted for baseline value and the randomization stratification factors; Difference from Placebo = 10.02, 95% CI 2-sided [9.04 to 11.01]

3. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 36 at Pre-selected Sites
Description: Bone mineral density was assessed by dual x-ray absorptiometry.
Time Frame: Baseline and Month 36
Population: BMD Analysis Set: all participants with total hip BMD evaluable values at Baseline and Month 36
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change in BMD
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 237 | 231
Percent Change in BMD | -3.32 [-4.06 to -2.58] | 4.60 [3.85 to 5.35]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p < 0.0001, ANCOVA — The Hochberg procedure was used to control for multiplicity; [statistical method as in outcome 2, analysis 1]; Difference from Placebo = 7.92, 95% CI 2-sided [6.87 to 8.97]

4. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Month 36 at Pre-selected Sites
Description: Bone mineral density was assessed by dual x-ray absorptiometry.
Time Frame: Baseline and Month 36
Population: BMD Analysis Set: all participants with evaluable femoral neck BMD values at Baseline and Month 36
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change in BMD
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 238 | 231
Percent Change in BMD | -3.10 [-3.72 to -2.48] | 3.41 [2.78 to 4.04]
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p < 0.0001, ANCOVA — The Hochberg procedure was used to control for multiplicity; [statistical method as in outcome 2, analysis 1]; Difference from Placebo = 6.51, 95% CI 2-sided [5.62 to 7.39]

5. Secondary Outcome: Number of Participants With New Vertebral Fractures
Description: Assessment of vertebral fractures was performed by an expert radiologist at the central imaging center using a semiquantitative grading scale: Grade 1, 20% to 25% reduction in vertebral height (anterior, middle, or posterior); Grade 2, 25% to 40% reduction in height; Grade 3, greater than 40% reduction in height.
  A new vertebral fracture was defined as a fracture in a previously undeformed vertebrae including new compression fractures, defined as those compression fractures having a decrease in total anterior or posterior height of at least 25% from baseline. New vertebral fractures includes morphometric vertebral fractures identified from on study x-rays and clinical vertebral fractures confirmed by x-rays.
Time Frame: 36 months
Population: Vertebral Fracture Analysis Set: all participants with a Baseline and at least one post-baseline vertebral x-ray prior to or at Month 36
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 809 | 835
Participants | 49 | 27
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p = 0.0088, Regression, Logistic; Logistic regression model includes treatment groups as the independent variable and stratified by the randomization stratification factors; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.33 to 0.85] — Values < 1 for odds ratio favor denosumab

6. Secondary Outcome: Number of Participants With New or Worsening Vertebral Fractures
Description: Assessment of vertebral fractures was performed by an expert radiologist at the central imaging center using a semiquantitative grading scale: Grade 1, 20% to 25% reduction in vertebral height (anterior, middle, or posterior); Grade 2, 25% to 40% reduction in height; Grade 3, greater than 40% reduction in height.
  A new vertebral fracture was defined as a fracture in a previously undeformed vertebrae including new compression fractures, defined as those compression fractures having a decrease in total anterior or posterior height of at least 25% from baseline. New vertebral fractures includes morphometric vertebral fractures identified from on study x-rays and clinical vertebral fractures confirmed by x-rays. Worsening of pre-existing fractures was defined as an increase in fracture severity of at least 1 grade on the semiquantitative scale.
Time Frame: 36 months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 809 | 835
Participants | 55 | 31
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority or Other; p = 0.0070, Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.34 to 0.84] — Values < 1 for odds ratio favor denosumab

7. Secondary Outcome: Disease-free Survival (DFS)
Description: DFS was defined as the time interval from the randomization date to the date of first evidence of local or distant metastases, contra-lateral breast cancer, secondary carcinoma, or death from any cause (whichever occurred first). Participants last known to be alive, who did not experience recurrence of disease, were censored at their last contact date or at the data cut-off date whichever came first.
Time Frame: From randomization until the DFS data cut-off date of 15 September 2015; maximum time on main study at the cut-off was 102 months
Population: Full Analysis Set: all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 1709 | 1711
Days | NA [NA to NA] — Not reached due to the low number of events | NA [NA to NA] — Not reached due to the low number of events
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority; p = 0.0515, Cox Proportional Hazards Model; Stratified by randomization strata (hospital type, use of aromatase inhibitor, baseline lumbar spine BMD); Hazard Ratio (HR) = 0.816, 95% CI 2-sided [0.66 to 1.00] — From the Cox Proportional hazards model with treatment fitted as a covariate and stratified by randomization strata. A hazard ratio < 1.0 indicates a lower average event rate and a longer disease-free time for denosumab relative to placebo

8. Secondary Outcome: Bone Metastases-free Survival (BMFS)
Description: BMFS was defined as the time interval from randomization to first occurrence of bone metastasis or death from any cause, whichever comes first. Participants last known to be alive, who did not experience bone metastasis, were censored at their last assessment (i.e., bone scan) date or at the last contact date, whichever comes first.
Time Frame: From randomization until end of main study, maximum time on main study was 152 months
Population: Full Analysis Set: all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 1709 | 1711
Days | NA [NA to NA] — Not reached due to the low number of events. | NA [NA to NA] — Not reached due to the low number of events.
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority — Analysis of BMFS was conditional on the outcome of DFS due to hierarchical testing strategy, therefore p-value not reported; Hazard Ratio (HR) = 0.808, 95% CI 2-sided [0.654 to 0.997] — A hazard ratio < 1.0 indicates a lower average event rate and a longer bone metastases-free time for denosumab relative to placebo

9. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: Randomization until end of main study, maximum duration of main study was 152 months
Population: Full analysis set: all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Denosumab
Number analyzed (Participants) | 1709 | 1711
Days | NA [NA to NA] — Not reached due to the low number of events. | NA [NA to NA] — Not reached due to the low number of events.
Statistical Analysis 1: Comparison: Placebo vs Denosumab; Test type: Superiority — Analysis of OS was conditional on the outcome of DFS due to hierarchical testing strategy, therefore p-value not reported; Hazard Ratio (HR) = 0.802, 95% CI 2-sided [0.635 to 1.013] — A hazard ratio < 1.0 indicates a lower average event rate and a longer overall survival time for denosumab relative to placebo

ADVERSE EVENTS:
Time Frame: Double-blind (DB) phase: from 1st dose of study drug to 30 days after last dose; Open-label (OL) phase: from 1st dose of OL study drug to 30 days after last dose. Median duration of treatment in DB phase: Placebo 35.4 months and denosumab 35.5 months. Median duration of treatment in OL phase: 37 months
Description: All randomized participants who received >1 dose of treatment; participants were analyzed according to the actual treatment received in double-blind phase. 9 participants randomized to the placebo in the DB phase incorrectly received denosumab. Per protocol, only AEs of special interest and SAEs were collected in the open-label phase. MedDRA 17.1 used in double-blind phase and 24.0 in the open-label phase.
Groups:
- Double-blind Phase: Placebo: Participants received the matching placebo SC Q6M in the double-blind phase. All participants continued to receive an approved non-steroidal aromatase inhibitor therapy.
- Double-blind Phase: Denosumab: Participants received 60 mg denosumab SC Q6M in the double-blind phase. All participants continued to receive an approved non-steroidal aromatase inhibitor therapy.
- Open-label Phase: Placebo/Denosumab: Participants who received the matching placebo during the double-blind phase, who continued into the open-label phase where they received denosumab 60 mg SC Q6M for up to a maximum of 7 additional doses.
- Open-label Phase: Denosumab/Denosumab: Participants who received denosumab during the double-blind phase, who continued into the open-label phase where they received denosumab 60 mg SC Q6M for up to a maximum of 7 additional doses.
Arm/Group | Double-blind Phase: Placebo | Double-blind Phase: Denosumab | Open-label Phase: Placebo/Denosumab | Open-label Phase: Denosumab/Denosumab
Serious Adverse Events (participants affected / at risk) | 515/1690 | 521/1709 | 40/245 | 0/1
Other Adverse Events (participants affected / at risk) | 838/1690 | 882/1709 | 0/245 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: Placebo (N=1690) | Double-blind Phase: Denosumab (N=1709) | Open-label Phase: Placebo/Denosumab (N=245) | Open-label Phase: Denosumab/Denosumab (N=1)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 3 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 4 | 5 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 2 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 2 | 4 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 11 | 14 | 3 | 0
Atrial flutter (Cardiac disorders) | 2 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 3 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 8 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 2 | 1 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 2 | 0 | 0
Coronary artery disease (Cardiac disorders) | 11 | 10 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 2 | 0 | 0
Myocardial infarction (Cardiac disorders) | 5 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Gene mutation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Ear canal stenosis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 10 | 9 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 4 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 0 | 0 | 0
Goitre (Endocrine disorders) | 12 | 21 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 2 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Blepharochalasis (Eye disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 28 | 16 | 2 | 0
Cataract cortical (Eye disorders) | 1 | 1 | 0 | 0
Cataract nuclear (Eye disorders) | 1 | 3 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0 | 0
Exfoliation glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 1 | 0 | 0 | 0
Macular fibrosis (Eye disorders) | 1 | 0 | 0 | 0
Open angle glaucoma (Eye disorders) | 0 | 1 | 0 | 0
Retinal degeneration (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 2 | 0 | 0
Retinal tear (Eye disorders) | 0 | 2 | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Vitreous opacities (Eye disorders) | 1 | 0 | 0 | 0
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Colon dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 7 | 7 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 4 | 8 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Oesophageal motility disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Painful defaecation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 3 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Peritoneal necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 2 | 4 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 8 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 3 | 2 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 9 | 14 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 2 | 0 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 5 | 0 | 0
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Borrelia infection (Infections and infestations) | 2 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 1 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 6 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 2 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 2 | 0 | 0 | 0
Device related infection (Infections and infestations) | 3 | 2 | 0 | 0
Diverticulitis (Infections and infestations) | 9 | 9 | 3 | 0
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0
Erysipelas (Infections and infestations) | 10 | 15 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Eye infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 2 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 6 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Haematoma infection (Infections and infestations) | 2 | 0 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 3 | 2 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 1 | 0 | 0
Incision site abscess (Infections and infestations) | 0 | 1 | 0 | 0
Infected seroma (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Joint abscess (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 1 | 0
Mastitis (Infections and infestations) | 1 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 3 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 9 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 2 | 0 | 0
Postoperative wound infection (Infections and infestations) | 2 | 0 | 0 | 0
Psoas abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 2 | 3 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 4 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Salpingitis (Infections and infestations) | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 4 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 3 | 6 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 9 | 7 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Bursa injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 5 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 6 | 4 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Haemodilution (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 3 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 24 | 23 | 0 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Radiation alveolitis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 5 | 2 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Splenic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 0
Suture rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood pressure abnormal (Investigations) | 0 | 1 | 0 | 0
Colonoscopy (Investigations) | 0 | 1 | 0 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 0 | 0
Mammogram abnormal (Investigations) | 0 | 1 | 0 | 0
Pulmonary arterial pressure increased (Investigations) | 1 | 0 | 0 | 0
Smear cervix abnormal (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Insulin resistance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 10 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 6 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 12 | 13 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 15 | 14 | 5 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Ligament disorder (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 6 | 8 | 1 | 0
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 59 | 62 | 2 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 4 | 9 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 6 | 2 | 0 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Benign lymph node neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3 | 1 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Contralateral breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Inflammatory myofibroblastic tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lobular breast carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Mediastinum neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Oral fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4 | 0 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0
Transitional cell carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Acoustic neuritis (Nervous system disorders) | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 1 | 0 | 0
Amnestic disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 2 | 0 | 0 | 0
Carotid artery disease (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 2 | 1 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 13 | 14 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 9 | 6 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Cervical myelopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 2 | 3 | 0 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0 | 0
Diabetic coma (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Drop attacks (Nervous system disorders) | 0 | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Facial neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 2 | 0 | 0
Medication overuse headache (Nervous system disorders) | 0 | 1 | 0 | 0
Meralgia paraesthetica (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Monoplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Morton's neuralgia (Nervous system disorders) | 1 | 1 | 0 | 0
Motor neurone disease (Nervous system disorders) | 1 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Radicular syndrome (Nervous system disorders) | 1 | 2 | 0 | 0
Sciatica (Nervous system disorders) | 4 | 7 | 1 | 0
Senile dementia (Nervous system disorders) | 0 | 1 | 0 | 0
Small fibre neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 4 | 6 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 3 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 2 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Burnout syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 8 | 8 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 2 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychosomatic disease (Psychiatric disorders) | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 1 | 0 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 1 | 0 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 2 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 4 | 0 | 0
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 2 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Adnexa uteri cyst (Reproductive system and breast disorders) | 0 | 2 | 0 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast calcifications (Reproductive system and breast disorders) | 4 | 4 | 0 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Breast discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast disorder (Reproductive system and breast disorders) | 6 | 1 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Breast fibrosis (Reproductive system and breast disorders) | 3 | 2 | 0 | 0
Breast haematoma (Reproductive system and breast disorders) | 2 | 1 | 0 | 0
Breast necrosis (Reproductive system and breast disorders) | 1 | 3 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 4 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 3 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 2 | 3 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 3 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 7 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 3 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Uterine adhesions (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 3 | 4 | 0 | 0
Uterine prolapse (Reproductive system and breast disorders) | 2 | 1 | 0 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 2 | 2 | 0 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 12 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 0
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Acquired epidermolysis bullosa (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Breast reconstruction (Surgical and medical procedures) | 0 | 1 | 0 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Intraocular lens implant (Surgical and medical procedures) | 0 | 1 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Mastectomy (Surgical and medical procedures) | 3 | 1 | 0 | 0
Oophorectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Prophylaxis (Surgical and medical procedures) | 0 | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 0
Arterial stenosis (Vascular disorders) | 2 | 0 | 0 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 4 | 3 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 2 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 2 | 0 | 0
Haematoma (Vascular disorders) | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 6 | 5 | 1 | 0
Hypertensive crisis (Vascular disorders) | 14 | 10 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 2 | 5 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 3 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 1 | 3 | 0 | 0
Peripheral venous disease (Vascular disorders) | 4 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Subclavian steal syndrome (Vascular disorders) | 1 | 0 | 0 | 0
Temporal arteritis (Vascular disorders) | 0 | 2 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 10 | 12 | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 2 | 0 | 0
Chest pain (General disorders) | 7 | 4 | 1 | 0
Cyst (General disorders) | 1 | 1 | 0 | 0
Device connection issue (General disorders) | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 4 | 3 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0
Fat necrosis (General disorders) | 1 | 2 | 0 | 0
Fibrosis (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 3 | 0 | 0
Granuloma (General disorders) | 0 | 1 | 0 | 0
Hyperplasia (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 4 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0
Medical device complication (General disorders) | 1 | 1 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 0 | 0
Oedema peripheral (General disorders) | 2 | 3 | 0 | 0
Pain (General disorders) | 2 | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia legionella (Infections and infestations) | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Paresis (Nervous system disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hydrometra (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-blind Phase: Placebo (N=1690) | Double-blind Phase: Denosumab (N=1709) | Open-label Phase: Placebo/Denosumab (N=245) | Open-label Phase: Denosumab/Denosumab (N=1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 446 | 441 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 146 | 151 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 111 | 139 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 61 | 89 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 85 | 107 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 73 | 89 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 86 | 78 | 0 | 0
Hot flush (Vascular disorders) | 234 | 270 | 0 | 0
Hypertension (Vascular disorders) | 94 | 111 | 0 | 0
Fatigue (General disorders) | 100 | 109 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT00556374/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT00556374/SAP_001.pdf